CLINICAL TRIAL: NCT03035396
Title: Clinical Performance of the Diassess Influenza A and B Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diassess Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DIA 01A-CLI-002
Record Dates: First submitted 2017-01-20; First posted 2017-01-30 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Influenza, Human; Influenza; Flu
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diassess Influenza A and B Test (Experimental)
  Interventions: Device: Diassess Influenza A and B Test

INTERVENTIONS:
Device: Diassess Influenza A and B Test

SUMMARY:
The primary objective of this study is device feasibility of the Diassess Influenza A and B Test

ELIGIBILITY:
Inclusion Criteria:

* Subject currently has a fever (≥37.8°C/100°F), or self-reports having had or is currently treating a fever ≥37.8°C/100°F with onset within the previous 72 hrs
* Subject has at least one additional flu-like symptom including fever or feeling feverish/chills, runny or stuffy nose, muscle or body aches, fatigue (very tired), sore throat, headaches, or cough

Exclusion Criteria:

* Subject received nasal vaccine (e.g. FluMist) within the past 10 days
* Subject has been taking or took any antivirals for influenza in the past 30 days
* Subject enrolled in any drug trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Diassess test measurement agreement with Polymerase Chain Reaction (PCR) | One (1) patient visit which is a time frame of one (1) hour

CONTACTS AND LOCATIONS:
Overall Officials: Carol Chen, PhD, Study Director — Diassess Inc.
Locations (1):
- University Health Care Center, Syracuse, New York, United States